CLINICAL TRIAL: NCT04867031
Title: Impact of the Food Matrix on Iodine Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: British Broadcasting Corporation (Industry)
Responsible Party: Principal Investigator, Emilie Combet, Senior Lecturer in Nutrition, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200160161
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Iodine Bioavailability
Keywords: iodine; bioavailability; seaweed; milk; fish
MeSH Terms: interventions — Milk; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White fish (cod) (Experimental): Participants will consume 1 portion (~130g) of white fish (Bird's Eye Inspirations Cod Fillets with Tomato & Rosemary), providing approximately 140µg of iodine, alongside 452mL of water. Urine will be collected for 36 hours following test food consumption.
  Interventions: Dietary Supplement: Fish
- Semi-skimmed milk (Experimental): Participants will consume 1 portion (~450mL) of milk (Tesco UHT Semi-Skimmed), providing approximately 140µg of iodine, alongside 452mL of water. Urine will be collected for 36 hours following test food consumption.
  Interventions: Dietary Supplement: Milk
- Dried seaweed sheets (Experimental): Participants will consume 1 portion (~6g) of dried seaweed sheets (Itsu Crispy Seaweed Thins), providing approximately 140µg of iodine, alongside 452mL of water. Urine will be collected for 36 hours following test food consumption.
  Interventions: Dietary Supplement: Seaweed

INTERVENTIONS:
Dietary Supplement: Milk — One portion of semi-skimmed cow's milk (approx. 450mL), providing ~140µg of iodine.
  Arms: Semi-skimmed milk
Dietary Supplement: Fish — One portion of cod (approx. 130g), providing ~140µg of iodine.
  Arms: White fish (cod)
Dietary Supplement: Seaweed — One portion of dried seaweed sheets (approx. 6g), providing ~140µg of iodine.
  Arms: Dried seaweed sheets

SUMMARY:
This study is a randomized crossover trial, lasting 12 days in total, which will assess the difference in iodine bioavailability (as a percentage of iodine consumed that is excreted in urine) from three iodine-rich foods; semi-skimmed milk, white fish, and dried seaweed sheets. Each of the three foods will provide approximately 140µg of iodine, and iodine excretion will be monitored for 36 hours following food ingestion via collection and analysis of urine.

DETAILED DESCRIPTION:
Iodine insufficiency is one of the three key micronutrient deficiencies highlighted as major public health issues by the World Health Organisation, and recent evidence indicates that the UK is now iodine deficient. Iodine deficiency represents a particular threat for women of child-bearing age, unborn infants and young children, as iodine is essential to synthesise the thyroid hormones, which are involved in key metabolic function including fetal brain development. Maternal iodine deficiency and the resulting changes in thyroid function has been associated with adverse pregnancy outcomes including spontaneous miscarriage, fetal distress and death, preterm delivery, low birth weight and impaired neuropsychological development, with significant impact on later life development and quality of life.

There is no iodine fortification programme in the United Kingdom, and despite worldwide efforts to tackle iodine deficiency and associated disorders via iodine supplementation and food-fortification (of salt mainly), consumption of supplements in the UK is virtually non-existent, with iodised salt used by less than 5%.

In the UK, the main dietary sources of iodine are dairy and sea-foods. Our previous studies have shown that seaweed intake can increase the iodine status of women with diets habitually low in iodine. Reduced bioavailability of iodine from the seaweed matrix, which could have implications for dietary recommendations.

This study address the influence of the food matrix on iodine bioavailability, in the context of food guidelines and assessment of the iodine status.

This project is in collaboration with the British Broadcast Corporation (BBC).

The study design is a crossover randomised trial - to last 9 days, plus three days pre-trial washout [total 12 days] - with 3 arms:

1. fish arm: portion equivalent to 140 µg iodine, approx. 130g.
2. milk arm: portion equivalent to 140 µg iodine, approx. 450mL.
3. seaweed arm: portion equivalent to 140 µg iodine, approx. 6g.

Each arm will be separated by two washout days, and participants will follow a low iodine diet (avoiding dairy, and all seafood) throughout the study, as well as three days prior to the first arm. Iodine levels will be monitored in urine collected during the 12 hours preceding and 36 hours following the meal. Urine will be collected in time fractions

A parallel design study showed that 56% (SD 20%) of a dose of potassium iodide is excreted after 24hours, compared to 36% (SD 13%) when the same dose comes from seaweed. In order to detect a similar difference, a sample of at least 13 participants is required (n=19 to allow for 30% attrition).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male or female
* Aged 18-48
* Signed informed consent

Exclusion Criteria:

* Pregnancy and lactation
* Past and present thyroid conditions
* Diseases of the gastrointestinal tract
* Allergy to seafood or dairy
* Consumption of iodine supplements
* Currently taking medication (other than the contraceptive pill)
* Having a habitual diet very low in iodine (<1 portion of dairy per day, or < 1 portion of fish per week)

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Iodine concentration in urine (µg/L) | 36 hours (fractions: 1-2, 2-3, 3-5, 5-7, 7-12, 12-24, 24-36 hours)
  Measured using the Sandell-Kolthoff method

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Combet, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Section of Human Nutrition, University of Glasgow, Glasgow, North Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided